CLINICAL TRIAL: NCT02012478
Title: The Impact of a Motivational Interviewing (MI) Informed Text Messaging (SMS) Program Tailored to Level of Patient Activation on Glycemic Control in a Population of Poorly Controlled Diabetic Patients.
Brief Title: Using a Motivational Interviewing (MI) Informed Text Messaging Program to Lower Blood Sugar in Diabetic Patients.
Acronym: MI-SMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Center for Healthcare Improvement and Patient Safety (Unknown); Leonard Davis Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 817790
Record Dates: First submitted 2013-12-10; First posted 2013-12-16 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No intervention (No Intervention): baseline session - with surveys and HbA1C only
- MI-informed SMS intervention (Experimental): Baseline session with surveys & HbA1C MI baseline session Technology tutorial Intervention x 3 months
  Interventions: Behavioral: MI- informed SMS program

INTERVENTIONS:
Behavioral: MI- informed SMS program
  Arms: MI-informed SMS intervention

SUMMARY:
Despite advances in medical therapy for diabetes, significant numbers of patients fail to achieve adequate blood glucose control. Diabetic patients who engage in more self-care behaviors have better glycemic control, as measured by HbA1C. Patient "activation", defined as the knowledge, skills, beliefs, and behaviors to manage a chronic disease, is key to the performance of these self-care behaviors.

There is a growing literature on diabetes behavioral change interventions; however interventions are often developed and implemented without consideration of patients readiness to engage in lifestyle changes. Additionally, patient-tailored interventions require intensive clinical and financial resources, making them difficult to integrate into clinical practice. Mobile text messaging (SMS) programs have been successfully used to promote smoking cessation, alcohol cessation, and weight loss in diverse patient populations. SMS interventions for diabetes have also been developed, but they have been designed primarily to provide feedback on blood glucose management, rather than to motivate behavioral change. The few studies that included motivational content as a primary feature, did not tailor their intervention to a patient's readiness for change or rigorously describe their motivational intervention, and show limited efficacy.

To address these concerns, we will perform a three-month randomized controlled pilot study to develop and test a Motivational Interviewing (MI)-informed SMS intervention tailored to patient level of activation for patients with poorly controlled type II diabetes.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* type II diabetes
* poorly controlled diabetes (HbA1C >8 x 2 measurements, with goal < 8)

Exclusion Criteria:

* pregnancy
* non-English speaking or reading

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
hemoglobin A1C | three months

SECONDARY OUTCOMES:
PAM scale | 3 months

OTHER OUTCOMES:
Summary of Diabetes Self-Care Activities | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Judith Long, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Hospital, Philadelphia, Pennsylvania, United States